CLINICAL TRIAL: NCT05356468
Title: Effects of Additional Pain Neuroscience Education (Pne) With Therapeutic Exercises on Pain Intensity in Patients With Lumbar Radiculopathy
Brief Title: PNE With Therapeutic Exercises on Pain Intensity in Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01231 Hira hassan
Record Dates: First submitted 2022-04-28; First posted 2022-05-02 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured pain neuroscience education (Experimental): Pain neuroscience education will be given to both groups. Group A will receive Structured Pain Neuroscience Education along with therapeutic , balance exercises and Postural training.
  Interventions: Other: Structured pain neuroscience education
- Conventional treatment (Active Comparator): Group B will receive Pain Neuroscience Education along with therapeutic, balance exercises. The treatment will continue for 6 weeks. Three sessions will be given in a week. Assessment would be done on baseline and at the end of every third week.
  Each session will be of 45 minutes. 15min electrotherapy, 15 min conventional treatment, 15 min PNE education.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Structured pain neuroscience education — Structured pain neuroscience
  * Neurophysiology of pain
  * The PNE occurred with the use of pictures, examples, metaphors and drawings as needed
  * Metaphor Alarm system: Your nerves working like an alarm system to protect you.
  * BOOKLET Consist of education about pain neurophysiology.(31)
  * Steps of booklet :
    1. Extract content
    2. English to Urdu translation
    3. Content Validity
    4. Expert Panel review by Physiotherapists
    5. Content validity Analysis review(Focus Group)
    6. Pilot study 4 to 5 patients
    7. Content improved (PNE) and Finalized
    8. After Analysis RCT
  Arms: Structured pain neuroscience education
Other: Conventional Treatment — ELECTROTHERAPY MODALTIES-15 min
  * IFC (interferential current)IFC will be administered using following parameters: 80-150 watts, 4000 Hz, sweep on, 16.0-17.0 CV(26)
  * Hot pack(27)
  Therapeutic exercises
  * Strengthening (Back extensors, quadriceps, hamstring and VMO, gluteus maximums, gluteus medius, transverse abdominis.
  * Stretching hamstring and, calf stretching. Soft tissue mobilization(5) McKenzie based exercises(28) BALANCE EXERCISES
  * Single Leg Stance (static balance) Patient is instructed to stand on one leg,close his/her eyes and maintain this position as long as they could.
  * Tandem gait (dynamic balance) patient is instructed to walk a total of 5 laps on a 2-meter-long line with the heel of the front foot touching the fingertip of the back foot.(29)
  POSTURAL TRAINING
  * good posture when sitting standing and while driving
  * Avoid weight lifting
  * Avoid too much bed rest
  * Sit in firm places. (30)
  Arms: Conventional treatment

SUMMARY:
There is lack of structured pain neuroscience education in patients with lumber radiculopathy. Previously researches were done on pain neuroscience education before surgery of lumber radiculopathy. However this study will provide structured educational plan about pain neuroscience education along with therapeutic exercises to positively influence pain knowledge, dysfunction, and fear avoidance, limitation in movement and healthcare utilization in patients who have diagnosed with lumbar radiculopathy and don't want to undergo surgery.

DETAILED DESCRIPTION:
Radicular pain or radiculopathy, defined as spinal nerve root dysfunction causing dermatomal discomfort and paresthesia's, myotome weakness, and/or reduced deep tendon reflexes, is frequently associated with axial spine pain. It affects both men and women and is believed to impact 3 to 5 percent of the population. Radiculopathy is pain that radiates down the legs and is described as electric, burning, and acute pain. Radiculopathy is most caused by irritation of a specific nerve, which can occur anywhere along the nerve and is most often caused by a compressive force. It could be caused by bulging or herniated discs, facet or ligamentous hypertrophy, spondylolisthesis, or even neoplastic or infectious diseases.

LR is the second leading cause of disability according to a research published by Global Burden of Disease (GBD).Pain neuroscience education (PNE), also known as therapeutic neuroscience education (TNE), is a series of instructional sessions for patients that cover the neurobiology and neurophysiology of pain, as well as how the nervous system processes pain. PNE alters the way a patient perceives pain at first. For example, a patient may have assumed that damaged tissues were the source of their pain; yet, after learning more about pain neurophysiology, the patient realises that pain may not accurately reflect tissue health and instead be caused by extra-sensitive nerves.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lumbar radiculopathy ( disc bulge , disc herniation , lumbar stenosis, disk dehydration(13)
* Medication. (Patient already on prescriptions, using medicines)
* Duration of low back pain as the main symptom for at least 3 months

Exclusion Criteria:

* The presence of chronic-pain-related conditions (e.g. fibromyalgia, chronic fatigue syndrome.)
* Pregnancy
* Patients on treatment with alternative therapies.
* Patients with associated pathologies that make it impossible to perform a physical exercise program (myopathies, neurological diseases with significant impairment of functionality

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Change From Baseline in Pain Scores on the Numeric Pain Rating Scale to 4 weeks till 8 Weeks
  The NPRS is used to measure pain intensity, in which patients are asked to select a number (from 0-10) to represent their pain severity.Change from Baseline , to 4Weeks, till 8 weeks
Time Up and Go Test(TUG) | Change From Baseline in balance Scores on the Time Up and Go Test(TUG) to 4 weeks till 8 Weeks.
  Timed up and go test (TUG) was used for measuring the time needed by the participants to stand up from the chair, walk 3 m to a red marker, and return to the starting position on the chair. Change from Baseline , balance and fall prevention to 4Weeks, 8 weeks
Oswestry Disability Index | Change From Baseline in disability Scores on Oswestry Disability Index to 4 weeks till 8 Weeks.
  Change from Baseline , to 4Weeks, to 8 weeks
Fear avoidance belief questionnaire | Change From Baseline in fear Scores on Fear avoidance belief questionnaire to 4 weeks till 8 weeks.
  Fear avoidance belief questionnaire he FABQ comprises two subscales; one measures the potential influence of fear-avoidance beliefs on general physical activity Change from Baseline , to 4Weeks, to 8 weeks
Beck Depression Inventory | Change From Baseline in depression Scores on Beck Depression Inventory to 4 weeks till 8 weeks
  Beck Depression Inventory (BDI) is a 21-item self-reporting questionnaire for evaluating the severity of depression in normal and psychiatric populations. Change from Baseline , to 4Weeks, to 8 weeks
The Pittsburgh Sleep Quality Index | Change From Baseline in sleep quality Scores to 4 weeks till 8 weeks.
  The PSQI is a self-rating questionnaire resulting in a global score between 0 and 21 which consist of seven sub scores. Change from Baseline , to 4Weeks, to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah college of Rehabilitation and Allied Health sciences Islamabad
Locations (1):
- Misbah Ghous, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No